CLINICAL TRIAL: NCT00005627
Title: A Phase I Study of Estramustine, Taxotere and Carboplatin (ETP) in Patients With Horomone Refractory Prostate Cancer
Brief Title: Estramustine, Docetaxel, and Carboplatin in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: DFCI-98238; CDR0000067775 (Registry Identifier: PDQ (Physician Data Query)); RP-DFCI-98238; NCI-G00-1779
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2003-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Docetaxel; Estramustine

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel
Drug: estramustine phosphate sodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of estramustine, docetaxel, and carboplatin in treating patients who have prostate cancer that has not responded to hormonal therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of weekly docetaxel when combined with carboplatin and estramustine in patients with hormone refractory prostate cancer.
* Determine the safety and efficacy of this regimen in this patient population.

OUTLINE: This is a dose escalation study of docetaxel.

Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV over 1 hour on day 2 of weeks 1-3. Patients also receive carboplatin IV over 1 hour on day 2 of week 1 only. Treatment continues every 28 days for up to 6 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-5 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 5 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Disease progression following androgen ablation therapy (hormonal or surgical) by either:

  * Increase in the product of bidimensional diameters of 1 or more radiographically documented sites of measurable disease OR
  * Two consecutive increases in PSA documented over a previous reference value

    * First increase in PSA should occur a minimum of 1 week from the reference value and be confirmed
    * First PSA value is less than the previous value, then patient is eligible provided next PSA is greater than the second PSA
* Testosterone levels documented in the castrate range (i.e., less than 30 ng/mL)

PATIENT CHARACTERISTICS:

Age:

* 18 to 85

Performance status:

* CALGB 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin normal
* SGOT no greater than 2.5 times upper limit of normal (ULN) if alkaline phosphatase normal OR
* Alkaline phosphatase no greater than 4 times ULN if SGOT normal OR
* SGOT no greater than 1.5 times ULN and alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within past year
* No significant change in anginal pattern within past 6 months
* No New York Heart Association class II-IV heart disease
* No deep venous thrombosis within past year

Other:

* No significant peripheral neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior chemotherapy allowed except taxanes or platinum derivatives

Endocrine therapy:

* See Disease Characteristics
* At least 4 weeks since prior antiandrogens

Radiotherapy:

* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Oh, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Oh WK, Hagmann E, Manola J, George DJ, Gilligan TD, Jacobson JO, Smith MR, Kaufman DS, Kantoff PW. A phase I study of estramustine, weekly docetaxel, and carboplatin chemotherapy in patients with hormone-refractory prostate cancer. Clin Cancer Res. 2005 Jan 1;11(1):284-9. PMID 15671557